CLINICAL TRIAL: NCT03470883
Title: Predictive Factors for Failure or Success of Endoscopic Treatment of Superficial Colorectal Tumors
Acronym: REC
Status: Completed | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: REC-IPC 2017-035
Record Dates: First submitted 2018-03-13; First posted 2018-03-20 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-03

CONDITIONS: Superficial Colorectal Tumors
Keywords: endoscopic resection; colorectal adenomas; Colorectal adenocarcinomas

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- endoscopic resection of a colorectal lesion: Patient having undergone endoscopic resection of a colorectal lesion stage 4 or 5 of the modified Vienna classification during the last 5 years at the institute.
  Interventions: Other: Evaluation of the long-term complete remission rate (> 12 months)

INTERVENTIONS:
Other: Evaluation of the long-term complete remission rate (> 12 months) — Evaluation of the long-term complete remission rate (> 12 months)

SUMMARY:
To evaluate the long-term complete remission rate (> 12 months) after endoscopic treatment of early neoplastic colorectal lesions.

DETAILED DESCRIPTION:
Intra-mucous colorectal neoplasia lesions (or even with minimal mucosal infiltration), formerly treated surgically, are increasingly treated endoscopically.

The IPC as a center for interventional endoscopy has been taking care of these lesions for several years.

Resection techniques have diversified since the 2000s (polypectomy, monobloc or piecemeal mucosectomy, submucosal dissection ... etc) and the endoscopy team has developed its various techniques within the institute ; Practice has evolved and has not been studied or evaluated in recent years. The purpose of this study is to evaluate practices and to compare results with the literature, and to identify predictive factors for the failure or success of endoscopic treatment of these early neoplastic lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patient having undergone endoscopic resection of a colorectal lesion stage 4 or 5 of the modified Vienna classification during the last 5 years at the institute.

Exclusion Criteria:

* Adenomas with low grade dysplasia
* Endoscopic control not available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient having undergone endoscopic resection of a colorectal lesion stage 4 or 5 of the modified Vienna classification
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-11-02 (Actual)

PRIMARY OUTCOMES:
Complete long-term remission (> 12 months) | 13 months
  Evaluation of the long-term complete remission rate (> 12 months)

SECONDARY OUTCOMES:
Absence of residual lesion on early control (3 to 6 months) | 3 to 6 months
  Medium-term response rate (3 to 6 months)
Rates of medium and long-term recurrence | 13 months
  Recurrence rate in the medium and long term
Management of medium and long-term recurrence | 13 months
  Management of recurrence (endoscopic revision or surgery)
Morbidity and mortality rates | 13 months
  Morbidity and mortality rate of endoscopic resection
Lymph node or visceral metastatic evolution rate | 13 months
  Rate of pejorative lymph node or metastatic evolution (especially for lesions with microinfiltration of the submucosa)
Endoscopic description and anatomopathological results | 1 day
  Endoscopic and / or anatomopathological predictive factors of success (complete long-term remission)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe RATONE, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli Calmettes, Marseille, Bouches Du Rhone, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dixon MF. Gastrointestinal epithelial neoplasia: Vienna revisited. Gut. 2002 Jul;51(1):130-1. doi: 10.1136/gut.51.1.130. PMID 12077106
- [Background] Repici A, Pellicano R, Strangio G, Danese S, Fagoonee S, Malesci A. Endoscopic mucosal resection for early colorectal neoplasia: pathologic basis, procedures, and outcomes. Dis Colon Rectum. 2009 Aug;52(8):1502-15. doi: 10.1007/DCR.0b013e3181a74d9b. PMID 19617768
- [Background] Moss A, Williams SJ, Hourigan LF, Brown G, Tam W, Singh R, Zanati S, Burgess NG, Sonson R, Byth K, Bourke MJ. Long-term adenoma recurrence following wide-field endoscopic mucosal resection (WF-EMR) for advanced colonic mucosal neoplasia is infrequent: results and risk factors in 1000 cases from the Australian Colonic EMR (ACE) study. Gut. 2015 Jan;64(1):57-65. doi: 10.1136/gutjnl-2013-305516. Epub 2014 Jul 1. PMID 24986245
- [Result] Ferlitsch M, Moss A, Hassan C, Bhandari P, Dumonceau JM, Paspatis G, Jover R, Langner C, Bronzwaer M, Nalankilli K, Fockens P, Hazzan R, Gralnek IM, Gschwantler M, Waldmann E, Jeschek P, Penz D, Heresbach D, Moons L, Lemmers A, Paraskeva K, Pohl J, Ponchon T, Regula J, Repici A, Rutter MD, Burgess NG, Bourke MJ. Colorectal polypectomy and endoscopic mucosal resection (EMR): European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline. Endoscopy. 2017 Mar;49(3):270-297. doi: 10.1055/s-0043-102569. Epub 2017 Feb 17. PMID 28212588
- [Result] Belderbos TD, Leenders M, Moons LM, Siersema PD. Local recurrence after endoscopic mucosal resection of nonpedunculated colorectal lesions: systematic review and meta-analysis. Endoscopy. 2014 May;46(5):388-402. doi: 10.1055/s-0034-1364970. Epub 2014 Mar 26. PMID 24671869